CLINICAL TRIAL: NCT02930070
Title: Diagnostic Accuracy of qSOFA Score for the Diagnosis of Sepsis in General Wards: a Single Center Cohort Study
Brief Title: qSOFA in General Wards: the Accuracy in Diagnosis of Sepsis
Acronym: qSOFAGAUGE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: qSOFA GAUGE
Record Dates: First submitted 2016-10-09; First posted 2016-10-11 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Sepsis
Keywords: sepsis; qSOFA; SOFA; diagnostic accuracy
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- qSOFA(+)SOFA(+): Infection patients who has a qSOFA>=2 and SOFA>=2 in a same day within 28 day of hospital stay.This group has the greatest priority in the competition of inclusion of groups.
- qSOFA(-)SOFA(+): Infection patients who has a qSOFA<2 and SOFA>=2 in a same day within 28 day of hospital stay.This group has the secondary priority in the competition of inclusion of groups.
- qSOFA(+)SOFA(-): Infection patients who has a qSOFA>=2 and SOFA<2 in a same day within 28 day of hospital stay.This group has the third priority in the competition of inclusion of groups.
- qSOFA(-)SOFA(-): Infection patients who has a qSOFA<2 and SOFA<2 in a same day within 28 day of hospital stay.This group has the least priority in the competition of inclusion of groups.

SUMMARY:
The new definition of sepsis (sepsis 3.0) restricts the early diagnosis of sepsis in general wards. Despite an alternative process by using a simplified qSOFA score, many patients may still be left out. Whether these patients matter or not is unknown. This prospective cohort includes patients from ten general wards with high incidence of infection during a consecutive half year, obtains qSOFA and SOFA score, follows up prognostic data, therefore to compare patients under different groups, eventually to evaluate the diagnostic accuracy of qSOFA score in diagnosis of sepsis.

DETAILED DESCRIPTION:
The sepsis, which is considered as multi-organ dysfunction induced by infection, is a one of leading causes of death in hospital. In 2016, the third international consensus has modified the definition of sepsis from infection with >=2 of systemic inflammatory response syndrome (SIRS) criteria to infection with >=2 of sequential organ failure assessment (SOFA) score. This new definition, which well reflects the organ dysfunction nature of sepsis, however makes it difficult to diagnose sepsis in general wards. An alternative of process was put forward to compensate this weakness. For each infection patient in general, access a quick SOFA (qSOFA), if it is above 2 score, then conduct laboratory examination to get a SOFA score. This process is helpful to find out sepsis, but undoubtedly leave out some patients who meet the SOFA criteria without qSOFA >=2. Besides, there are also some patients who has a qSOFA >=2 however do not meet the SOFA criteria. Whether those patients have better survival rate is unclear. This prospective cohort is aimed to compare prognosis of patients with different SOFA, qSOFA score, therefore access the diagnostic accuracy of qSOFA in the diagnosis of sepsis, eventually evaluate the feasibility of using qSOFA as a complete replacement of SOFA in general wards.

ELIGIBILITY:
Inclusion Criteria:

* Age>=18;

Exclusion Criteria:

* Hospital stay less than 24h just for chemotherapy,biotherapy or endoscopy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with infection in 10 selected general wards
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | 28 day
  the mortality within 28 day of hospital stay

SECONDARY OUTCOMES:
Duration of stay in the hospital | 28 day
  the duration of hospital stay with first 28 day
Organ dysfunctions | 28 day
  the detailed items of SOFA to reflect major organ dysfunctions

CONTACTS AND LOCATIONS:
Overall Officials: Li Weng, MD, Principal Investigator — Medical ICU, Peking Union Medical College Hospital
Locations (2):
- China (2):
  - Medical ICU,Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Result] Shankar-Hari M, Phillips GS, Levy ML, Seymour CW, Liu VX, Deutschman CS, Angus DC, Rubenfeld GD, Singer M; Sepsis Definitions Task Force. Developing a New Definition and Assessing New Clinical Criteria for Septic Shock: For the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):775-87. doi: 10.1001/jama.2016.0289. PMID 26903336
- [Result] Churpek MM, Zadravecz FJ, Winslow C, Howell MD, Edelson DP. Incidence and Prognostic Value of the Systemic Inflammatory Response Syndrome and Organ Dysfunctions in Ward Patients. Am J Respir Crit Care Med. 2015 Oct 15;192(8):958-64. doi: 10.1164/rccm.201502-0275OC. PMID 26158402
- [Derived] Luo J, Jiang W, Weng L, Peng J, Hu X, Wang C, Liu G, Huang H, Du B. Usefulness of qSOFA and SIRS scores for detection of incipient sepsis in general ward patients: A prospective cohort study. J Crit Care. 2019 Jun;51:13-18. doi: 10.1016/j.jcrc.2019.01.012. Epub 2019 Jan 18. PMID 30685579